CLINICAL TRIAL: NCT05323058
Title: The Use of Tulsi Extract for The Management of Oral Mucositis in Head & Neck Cancer Patients Undergoing Radiotherapy: A Randomized Clinical Trial
Brief Title: The Use of Tulsi Extract for The Management of Oral Mucositis in Head & Neck Cancer Patients Undergoing Radiotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karima AbdAllah Kamel, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tulsi in radiation mucositis
Record Dates: First submitted 2022-03-27; First posted 2022-04-12 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Stomatitis
Keywords: oral mucositis; tulsi extract; benzydamine hydrochloride; radiotherapy
MeSH Terms: conditions — Stomatitis | interventions — holy basil leaf extract; Benzydamine

STUDY DESIGN:
Intervention Model Description: Allocation ratio (1:1)
Who Masked: Participant, Investigator
Masking Description: The principal investigator and participant will be blinded as the treatment preparations will be identical in color, odor, and consistency and they will be placed in identical bottles
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tulsi extract (Experimental): 4% tulsi extract as intervention
  Interventions: Drug: tulsi extract
- benzydamine hydrochloride (Active Comparator): 0.15% benzydamine hydrochloride
  Interventions: Drug: Benzydamine Hydrochloride

INTERVENTIONS:
Drug: tulsi extract — 4% topical oral spray
  Arms: tulsi extract
Drug: Benzydamine Hydrochloride — 0.15% topical oral spray
  Arms: benzydamine hydrochloride

SUMMARY:
After signing the informed consent, the participant will be allocated to either intervention or control group, then each participant will use either 0.15% benzydamine (Comparator) or 4% tulsi (Intervention) four times a day and also once half an hour before each radiotherapy session.

DETAILED DESCRIPTION:
the primary outcome is the severity of oral mucositis will assess by Oral Mucositis Assessment Scale (OMAS) and secondary outcomes are pain will assess Numerical rating scale (NRS), Oral Assessment Guide (OAG), and Patient-Reported Oral Mucositis( PROMS scale) All outcomes will be recorded at baseline, and 8, 15 days

ELIGIBILITY:
Inclusion Criteria:

* Patients having clinical signs of radiotherapy-induced OM (WHO oral mucositis grading scale: Grade II, III, and IV)
* Patient should be able to read and/or understand and sign the consent form.

Exclusion Criteria:

1. Patients with HIV infections or hyperthyroidism.
2. Karnofsky performance status (KPS) less than 60%
3. Patients having an allergy to tulsi or benzydamine HCL
4. Patients who are pregnant and/or nursing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Severity of mucositis | up to 15 days
  Oral Mucositis Assessment Scale (OMAS)

SECONDARY OUTCOMES:
Pain and burning sensation | up to 15 days
  assess by numerical rating scale (NRS) (10 points scale)

OTHER OUTCOMES:
Oral Assessment Guide (OAG) | up to 15 days
  Assessment of patient speech, salivary function and quality, gingival health, swallowing, lips, and oral hygiene.
Patient-Reported Oral Mucositis( PROMS scale) | up to 15 days
  Quality of life

IPD SHARING:
Plan to Share IPD: No